CLINICAL TRIAL: NCT01630434
Title: Prospective, International, Multi-Center, Randomized Clinical Investigation of TransMedics Organ Care System (OCS LUNG) for Lung Preservation and Transplantation
Brief Title: International Randomized Study of the TransMedics Organ Care System (OCS Lung) for Lung Preservation and Transplantation
Acronym: INSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OCS-LUN-03-2010
Record Dates: First submitted 2012-06-25; First posted 2012-06-28 (Estimated); Results first posted 2022-07-07 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2016-05

CONDITIONS: Lung Preservation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OCS Lung (Treatment Group) (Experimental): The OCS Lung, which is a portable, integrated platform designed to maintain adult donor lungs in a normothermic state through continuous normothermic perfusion and ventilation, will be used to preserve and transport donor lungs.
  Interventions: Device: OCS Lung
- Cold flush and storage (Control Group) (Active Comparator): Donor lungs will be preserved using cold flush and storage (control group)
  Interventions: Device: Cold flush and storage

INTERVENTIONS:
Device: OCS Lung — OCS Lung will be used to preserve the donor lungs (Treatment Group).
  Arms: OCS Lung (Treatment Group)
Device: Cold flush and storage — Donor lungs will preserved using standard cold flush and storage
  Other Names: Commercially available cold preservation solution
  Arms: Cold flush and storage (Control Group)

SUMMARY:
A prospective, international, multi-center, randomized controlled trial comparing preservation of donor lungs using OCS-Lung perfusion device (Treatment Group) to cold flush and storage (Control Group).

ELIGIBILITY:
Inclusion Criteria:

* Registered primary double-lung transplant candidate
* Age > or equal to 18
* Signed: 1) written informed consent document and 2) authorization to use and disclose protected health information

Exclusion Criteria:

* Prior solid organ or bone marrow transplant
* Single lung recipient
* Multiple organ transplant recipient
* Chronic use of hemodialysis or diagnosis of chronic renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2011-11; Primary Completion 2014-09 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abbas Ardehali, MD, Study Director — Ronald Reagan Medical Center, UCLA; Dirk van Raemodonck, MD, Study Director — UZ Leuven, Belgium; Gregor Warnecke, MD, Study Director — Hannover Medical Center, Germany
Locations (21):
- United States (8):
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - University of California at Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Indiana University, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- St. Vincent's Hospital, Darlinghurst, New South Wales, Australia
- Hospitals Leuven, Leuven, Belgium
- University of Alberta, Edmonton, Alberta, Canada
- France (3):
  - University Hospitals of Marseille, Marseille
  - Groupe Hospitalier Hopitaux Universitaries, Paris
  - N.H.C Hospital Civil, Strasbourg
- Germany (3):
  - German Heart Institute Berlin, Berlin
  - Universitäres Herzzentrum Hamburg GmbH, Hamburg
  - Hannover Medical School, Hanover
- University of Padua, Padua, Italy
- University Puerta de Hierro Hospital, Madrid, Spain
- United Kingdom (2):
  - Papworth Hospital, Cambridge
  - Harefield Hospital, Middlesex

REFERENCES:
- [Derived] Warnecke G, Van Raemdonck D, Smith MA, Massard G, Kukreja J, Rea F, Loor G, De Robertis F, Nagendran J, Dhital KK, Moradiellos Diez FJ, Knosalla C, Bermudez CA, Tsui S, McCurry K, Wang IW, Deuse T, Leseche G, Thomas P, Tudorache I, Kuhn C, Avsar M, Wiegmann B, Sommer W, Neyrinck A, Schiavon M, Calabrese F, Santelmo N, Olland A, Falcoz PE, Simon AR, Varela A, Madsen JC, Hertz M, Haverich A, Ardehali A. Normothermic ex-vivo preservation with the portable Organ Care System Lung device for bilateral lung transplantation (INSPIRE): a randomised, open-label, non-inferiority, phase 3 study. Lancet Respir Med. 2018 May;6(5):357-367. doi: 10.1016/S2213-2600(18)30136-X. Epub 2018 Apr 9. PMID 29650408
- [Derived] Bozso S, Freed D, Nagendran J. Successful transplantation of extended criteria lungs after prolonged ex vivo lung perfusion performed on a portable device. Transpl Int. 2015 Feb;28(2):248-50. doi: 10.1111/tri.12474. Epub 2014 Oct 27. No abstract available. PMID 25284600

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OCS Lung (Treatment Group) | Cold Flush and Storage (Control Group)
Started (Intention-to-treat population) | 151 | 169
Safety Population | 150 | 169
Per Protocol Population | 141 | 165
Completed (Number of per protocol subjects that completed 24-month follow-up) | 121 | 139
Not Completed | 30 | 30
Not completed — Donor lungs turned down | 1 | 0
Not completed — Protocol Violation | 9 | 4
Not completed — Death | 20 | 26

BASELINE CHARACTERISTICS:
Population: Intent-to-treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | OCS Lung (Treatment Group) | Cold Flush and Storage (Control Group) | Total
Number analyzed (Participants) | 151 | 169 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] — Donor Age (years)
  years | 42.2 (14.4) | 40.2 (13.7) | 41.1 (14.1)
Age, Continuous [Mean (Standard Deviation); unit: years] — Recipient Age (years)
  years | 50.4 (13.1) | 50.0 (13.6) | 50.2 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Donor Sex (Male/Female)
  Participants
    Female | 72 | 67 | 139
    Male | 79 | 102 | 181
Sex: Female, Male [Count of Participants; unit: Participants] — Recipient Sex (Male/Female)
  Participants
    Female | 74 | 63 | 137
    Male | 77 | 106 | 183
Donor Smoking History in Past 6 Months [Count of Participants; unit: Participants] | 27 | 27 | 54
Final PaO2:FiO2 (mm Hg) [Mean (Standard Deviation); unit: mm Hg] | 438.5 (80.0) | 431.7 (73.8) | 434.9 (76.7)
Recipient Transplant Indication [Count of Participants; unit: Participants]
  COPD | 46 | 52 | 98
  Pulmonary Fibrosis | 49 | 57 | 106
  Cystic Fibrosis | 31 | 40 | 71
  Idiopathic Pulmonary Hypertension | 13 | 6 | 19
  Sarcoidosis | 4 | 8 | 12
  Other | 8 | 6 | 14
Recipient Lung Allocation Score [Mean (Standard Deviation); unit: score on a scale] — Recipient lung allocation score (LAS) is the value that determines a recipient's urgency on the waitlist. This score is assigned on a scale of 0 to 100, 0 being the least urgent and 100 being the most urgent recipient.
  score on a scale | 50.8 (20.9) | 47.9 (18.7) | 49.3 (19.8)
Recipient BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.2 (4.6) | 23.0 (4.1) | 23.1 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: A Composite of Patient Survival at Day 30 Post Transplantation, and Absence of International Society for Heart & Lung Transplantation (ISHLT) Primary Graft Dysfunction (PGD3) Grade 3 Within the First 72 Hours Post-transplantation.
Description: This composite is a single outcome measure. Primary graft dysfunction is graded on a scale of 0 to 3 according to the 2005 ISHLT PGD grading consensus. Grade 0 is considered the least severe and grade 3 is considered a more severe outcome.
Time Frame: Day 30 after transplantation
Measure: Count of Participants; unit: Participants
Groups:
- OCS Lung (Treatment Group) - Per Protocol; OCS Lung (Treatment Group) - ITT: The OCS Lung, which is a portable, integrated platform designed to maintain adult donor lungs in a normothermic state through continuous normothermic perfusion and ventilation, will be used to preserve and transport donor lungs.
  OCS Lung: OCS Lung will be used to preserve the donor lungs (Treatment Group).
- Cold Flush and Storage (Control Group) - Per Protocol; Cold Flush and Storage (Control Group) - ITT: Donor lungs will be preserved using cold flush and storage (control group)
  Cold flush and storage: Donor lungs will preserved using standard cold flush and storage
Arm/Group | OCS Lung (Treatment Group) - Per Protocol | Cold Flush and Storage (Control Group) - Per Protocol | OCS Lung (Treatment Group) - ITT | Cold Flush and Storage (Control Group) - ITT
Number analyzed (Participants) | 141 | 165 | 151 | 169
Participants | 112 | 116 | 112 | 119
Statistical Analysis 1: Comparison: OCS Lung (Treatment Group) - Per Protocol vs Cold Flush and Storage (Control Group) - Per Protocol; Test type: Non-Inferiority — The non-inferiority margin, which is here taken to be 0.04; p = 0.004, Wald Method; difference of proportion = -0.091, 95% CI 1-sided [upper limit -0.01]
Statistical Analysis 2: Comparison: OCS Lung (Treatment Group) - ITT vs Cold Flush and Storage (Control Group) - ITT; Test type: Non-Inferiority — The non-inferiority margin, which is here taken to be 0.04; p = 0.06, Wald Method; difference of proportion = -0.038, 95% CI 1-sided [upper limit 0.045]

2. Secondary Outcome: Participants With International Society for Heart & Lung Transplantation (ISHLT) PGD Grade 3 at 72 Hours Post-transplantation
Description: Primary graft dysfunction is graded on a scale of 0 to 3 according to the 2005 ISHLT PGD grading consensus. Grade 0 is considered the least severe and grade 3 is considered a more severe outcome.
Time Frame: 72 hours after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | OCS Lung (Treatment Group) - Per Protocol | Cold Flush and Storage (Control Group) - Per Protocol | OCS Lung (Treatment Group) - ITT | Cold Flush and Storage (Control Group) - ITT
Number analyzed (Participants) | 141 | 165 | 151 | 169
Participants | 3 | 6 | 7 | 7
Statistical Analysis 1: Comparison: OCS Lung (Treatment Group) - Per Protocol vs Cold Flush and Storage (Control Group) - Per Protocol; Test type: Non-Inferiority — The non-inferiority margin is 5%; p = 0.0003, Wald Method; Difference of proportions = -0.015, 95% CI 1-sided [upper limit 0.016]
Statistical Analysis 2: Comparison: OCS Lung (Treatment Group) - ITT vs Cold Flush and Storage (Control Group) - ITT; Test type: Non-Inferiority — The non-inferiority margin is 5%; p = 0.027, Wald Method; Difference of proportions = 0.006, 95% CI 1-sided [upper limit 0.044]

3. Secondary Outcome: Participants With ISHLT PGD Grade 2 or 3 at 72 Hours Post-transplantation
Description: as for outcome 2
Time Frame: 72 hours after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | OCS Lung (Treatment Group) - Per Protocol | Cold Flush and Storage (Control Group) - Per Protocol | OCS Lung (Treatment Group) - ITT | Cold Flush and Storage (Control Group) - ITT
Number analyzed (Participants) | 141 | 165 | 151 | 169
Participants | 16 | 13 | 22 | 14
Statistical Analysis 1: Comparison: OCS Lung (Treatment Group) - Per Protocol vs Cold Flush and Storage (Control Group) - Per Protocol; Test type: Non-Inferiority — The non-inferiority margin is 7.5%; p = 0.118, Wald Method; Difference of proportions = 0.035, 95% CI 1-sided [upper limit 0.091]
Statistical Analysis 2: Comparison: OCS Lung (Treatment Group) - ITT vs Cold Flush and Storage (Control Group) - ITT; Test type: Non-Inferiority — The non-inferiority margin is 7.5%; p = 0.389, Wald Method; Difference of proportions = 0.065, 95% CI 1-sided [upper limit 0.124]

4. Secondary Outcome: Patient Survival at Day 30
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | OCS Lung (Treatment Group) - Per Protocol | Cold Flush and Storage (Control Group) - Per Protocol | OCS Lung (Treatment Group) - ITT | Cold Flush and Storage (Control Group) - ITT
Number analyzed (Participants) | 141 | 165 | 151 | 169
Participants | 135 | 165 | 142 | 168
Statistical Analysis 1: Comparison: OCS Lung (Treatment Group) - Per Protocol vs Cold Flush and Storage (Control Group) - Per Protocol; Test type: Non-Inferiority — The non-inferiority margin is 4%; Difference of proportions = 0.043, 95% CI 1-sided [upper limit 0.071]
Statistical Analysis 2: Comparison: OCS Lung (Treatment Group) - ITT vs Cold Flush and Storage (Control Group) - ITT; Test type: Non-Inferiority — The non-inferiority margin is 4%; Difference of proportions = 0.054, 95% CI 1-sided [upper limit 0.087]

5. Other Pre Specified Outcome: Primary Safety Endpoint: Lung Graft-related Serious Adverse Events (LGRSAEs) Through 30-days Post-transplant Per Subject
Description: An LGRSAE event is defined as the occurrence of any of the following four categories of adverse events that are also serious; acute rejection, respiratory failure, bronchial anastomotic complication, and major pulmonary-related infection.
Time Frame: 30 days post-transplant
Population: This analysis was done on the safety population.
Measure: Mean (95% Confidence Interval); unit: events per participant
Arm/Group | OCS Lung (Treatment Group) | Cold Flush and Storage (Control Group)
Number analyzed (Participants) | 150 | 169
events per participant | 0.23 [0 to 0.47] | 0.28 [0 to 0.47]
Statistical Analysis 1: Comparison: OCS Lung (Treatment Group) vs Cold Flush and Storage (Control Group); Test type: Non-Inferiority — The non-inferiority margin is 0.7; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = -0.045, 95% CI 1-sided [upper limit 0.047]

6. Other Pre Specified Outcome: Long-term Survival: 24-month Survival
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | OCS Lung (Treatment Group) - Per Protocol | Cold Flush and Storage (Control Group) - Per Protocol | OCS Lung (Treatment Group) - ITT | Cold Flush and Storage (Control Group) - ITT
Number analyzed (Participants) | 141 | 165 | 151 | 169
Participants | 121 | 139 | 127 | 142

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 30 days post-transplant or through hospital discharge if longer than 30 days. All-cause mortality is reported through 24-months post transplant.
Description: The primary safety endpoint was lung graft-related serious adverse events within 30 days (acute rejection, respiratory failure, bronchial anastomotic complications, and major pulmonary-related infection).
Arm/Group | OCS Lung (Treatment Group) | Cold Flush and Storage (Control Group)
All-Cause Mortality (participants affected / at risk) | 24/151 | 27/169
Serious Adverse Events (participants affected / at risk) | 83/150 | 107/169
Other Adverse Events (participants affected / at risk) | 125/150 | 141/169
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OCS Lung (Treatment Group) (N=150) | Cold Flush and Storage (Control Group) (N=169)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 42 (54) | 51 (66)
Infections and infestations (Infections and infestations) | 31 (36) | 50 (65)
Cardiac disorders (Cardiac disorders) | 15 (20) | 15 (16)
Renal and urinary disorders (Renal and urinary disorders) | 11 (11) | 12 (12)
Vascular disorders (Vascular disorders) | 11 (14) | 7 (7)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 11 (11) | 9 (9)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2) | 12 (16)
Immune system disorders (Immune system disorders) | 6 (6) | 12 (12)
Nervous system disorders (Nervous system disorders) | 8 (9) | 7 (7)
General disorders and administration site conditions (General disorders) | 2 (2) | 5 (5)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 4 (4)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hepatobiliary disorders (Hepatobiliary disorders) | 0 (0) | 1 (2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Surgical and medical procedures (Surgical and medical procedures) | 2 (2) | 0 (0)
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Investigations (Investigations) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OCS Lung (Treatment Group) (N=150) | Cold Flush and Storage (Control Group) (N=169)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 56 (79) | 69 (95)
Infections and infestations (Infections and infestations) | 42 (52) | 54 (72)
Cardiac disorders (Cardiac disorders) | 33 (39) | 46 (48)
Renal and urinary disorders (Renal and urinary disorders) | 18 (18) | 25 (25)
Vascular disorders (Vascular disorders) | 18 (22) | 12 (12)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 17 (18) | 18 (18)
Gastrointestinal disorders (Gastrointestinal disorders) | 8 (8) | 18 (25)
Immune system disorders (Immune system disorders) | 22 (23) | 32 (36)
Nervous system disorders (Nervous system disorders) | 21 (22) | 14 (15)
General disorders and administration site conditions (General disorders) | 5 (7) | 9 (9)
Psychiatric disorders (Psychiatric disorders) | 7 (7) | 10 (10)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 4 (5) | 7 (7)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 7 (7) | 7 (8)
Hepatobiliary disorders (Hepatobiliary disorders) | 0 (0) | 1 (2)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Surgical and medical procedures (Surgical and medical procedures) | 2 (3) | 2 (2)
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Investigations (Investigations) | 5 (5) | 14 (15)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Endocrine disorders (Endocrine disorders) | 0 (0) | 2 (2)
Eye disorders (Eye disorders) | 2 (2) | 0 (0)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site shall have right to publish results. To balance this right with TransMedics' (TM) proprietary interests, site will submit manuscripts intended for publication for TM's review at least 60d prior to submission date. TM will complete its review within 60d of receipt. TM may request that site delete from its manuscripts any reference to TM confidential information and site shall promptly comply with such request. After 60d period, site will have right to publish manuscript, as amended by TM.